CLINICAL TRIAL: NCT05066984
Title: Evaluation of Structured, Multidisciplinary and Personalized Post-ICU Care on Physical and Psychological Functioning, and Quality of Life of Former ICU Patients
Brief Title: MONITOR-IC Post ICU Care Study
Acronym: MiCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch National Health Care Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13125
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Post ICU Syndrome
Keywords: post-ICU care; cost-effectiveness; QoL; PROMs

STUDY DESIGN:
Intervention Model Description: Multicenter stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- structured, multidisciplinary and personalized post-ICU care (Experimental): structured, multidisciplinary and personalized post-ICU care
  Interventions: Other: structured, multidisciplinary and personalized post-ICU care
- Ususal care (No Intervention): Usual care

INTERVENTIONS:
Other: structured, multidisciplinary and personalized post-ICU care — Structured, personalized and multidisciplinary post-ICU care tailored to patients' health problems initiated by ICU clinicians and coordinated by GPs.
  Arms: structured, multidisciplinary and personalized post-ICU care

SUMMARY:
* OBJECTIVE To evaluate the clinical effectiveness and cost effectiveness of structured, multidisciplinary and personalized post-ICU care versus usual care on physical and psychological functioning, and quality of life (QoL) of ICU survivors one and two years post-ICU.
* RESEARCH QUESTION What is the clinical- and cost effectiveness of structured, personalized post-ICU care versus usual care on physical and psychological functioning, and QoL of ICU survivors?
* HYPOTHESIS Structured, multidisciplinary, and personalized post-ICU care results in improved QoL of ICU survivors and is more cost effective compared to usual care.

DETAILED DESCRIPTION:
* OBJECTIVE To evaluate the clinical effectiveness and cost effectiveness of structured, multidisciplinary and personalized post-ICU care versus usual care on physical and psychological functioning, and quality of life (QoL) of ICU survivors one and two years post-ICU.
* RESEARCH QUESTION What is the clinical- and cost effectiveness of structured, personalized post-ICU care versus usual care on physical and psychological functioning, and QoL of ICU survivors?
* HYPOTHESIS Structured, multidisciplinary, and personalized post-ICU care results in improved QoL of ICU survivors and is more cost effective compared to usual care.
* STUDY POPULATION Adult patients at high risk of critical illness-associated morbidity post-ICU.
* INTERVENTION Structured, personalized and multidisciplinary post-ICU care tailored to patients' health problems initiated by ICU clinicians and coordinated by GPs.
* USUAL CARE / COMPARISON No or unstructured post-ICU care.
* OUTCOMES Primary: QoL and mental functioning 1-year post-ICU. Secondary: physical and cognitive functioning 1- and 2-year post-ICU, cost effectiveness and cost utility.
* FOLLOW-UP TIME One and two years post-ICU.
* STUDY DESIGN Stepped wedge cluster RCT in 5 hospitals.
* SAMPLE SIZE & DATA ANALYSIS 5 ICUs (11 patients/ICU/month, in total 770 intervention patients, and 1480 (active and historical) controls gives power of 87% to detect effect of 0.074 in EQ-5D (ICC 0.035; SD 0.26). Data will be analysed according to intention to treat principles, also per-protocol analyses will be performed.
* COST-EFFECTIVENESS ANALYSIS / BUDGET IMPACT ANALYSIS Comparison of 'cost per QALY' gained between patients in the intervention and control group. Decision analytical modelling will be used to calculate the average savings per patient; extrapolated to population level using a budget-holders perspective.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients at high risk of critical illness-associated morbidity post-ICU
* 18 years or older
* Patient or legal representative understands the Dutch language

Exclusion Criteria:

* Patients discharged from ICU/hospital direct to a nursing home
* Patients discharged from ICU/hospital direct to a medical or geriatric rehabilitation clinic
* Patients discharged for palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Individual's perception of their position in life assessed by the EuroQol-5 dimension (EQ5D) . | 1 year post-ICU
  Quality of life (QoL) assessed by the EQ5D at 1-year post-ICU.
Mental impairments assessed by the Hospital Anxiety and Depression Scale (HADS) | 1 year post-ICU
  Anxiety and depression (assessed by the HADS) at 1-year post-ICU.

SECONDARY OUTCOMES:
Physical functioning measured by fatigue assessed by the Checklist Individual Strength (CIS). | 1- and 2-year post-ICU
  Fatigue (CIS) Patients' level of frailty and vulnerability will be assed using the Clinical Frailty Score (CFS).
Physical functioning measured by frailty assessed by the Clinical Frailty Scale (CFS). | 1- and 2-year post-ICU
  Frailty (CFS) Patients' level of frailty and vulnerability will be assed using the Clinical Frailty Score (CFS).
Physical functioning measured by new physical complaints assessed by the number of new physical complaints. | 1- and 2-year post-ICU
  New physical complaints Patients' level of frailty and vulnerability will be assed using the Clinical Frailty Score (CFS).
Post traumatic stress disorder 1- and 2-year post-ICU assessed by the Impact of Event Scale-Revised (IES-R). | 1- and 2-year post-ICU
  Post traumatic stress disorder (IES-R)
Cognitive functioning 1- and 2-year post-ICU assessed by the 14-item Cognitive Failure Questionnaire (CFQ14). | 1- and 2-year post-ICU
  Cognitive functioning (CFQ14)
Social economic consequences measured by the novel question set designed by Griffiths et al. | 1- and 2-year post-ICU
  Social consequences and return to work will be measured using the novel question set designed by Griffiths et al to determine changes in family circumstances, socioeconomic stability and care requirements.
  (Griffiths J, Hatch RA, Bishop J, et al. An exploration of social and economic outcome and associated health-related quality of life after critical illness in general intensive care unit survivors: a 12-month follow-up study. Critical care. 2013;17(3):R100.)
Cost effectiveness measured by cost per Quality-Adjusted Life Years (QALY) | 1- and 2-year post-ICU
  A cost-effectiveness analysis will be carried out to evaluate whether the costs of structured, multidisciplinary and personalized post-ICU care weigh up to the benefits compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, PhD, Study Director — Radboud University Medical Center; Marieke Zegers, PhD, Study Director — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on reasonable request to the researchers.
Supporting Information: Study Protocol, ICF
Time Frame: After finalizing the final analysis in 2026 for a period of 5 years.
Access Criteria: Data will be shared on reasonable request to the researchers.

REFERENCES:
- [Derived] van Sleeuwen D, van de Laar FA, Simons K, van Bommel D, Burgers-Bonthuis D, Koeter J, Bisschops LLA, Vloet L, Brackel M, Teerenstra S, Adang E, van der Hoeven JG, Zegers M, van den Boogaard M. MiCare study, an evaluation of structured, multidisciplinary and personalised post-ICU care on physical and psychological functioning, and quality of life of former ICU patients: a study protocol of a stepped-wedge cluster randomised controlled trial. BMJ Open. 2022 Sep 15;12(9):e059634. doi: 10.1136/bmjopen-2021-059634. PMID 36109035